CLINICAL TRIAL: NCT01647672
Title: A Study to Assess the Efficacy and Safety With Albumin-bound Paclitaxel (Abraxane) in the TAC as Neoadjuvant Chemotherapy in the Treatment of Operable Breast Cancer
Brief Title: Efficacy and Safety With Albumin-bound Paclitaxel (Abraxane) in the TAC as Neoadjuvant Chemotherapy in Breast Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University (Other)
Responsible Party: Principal Investigator, Zhang jin, Professor, Tianjin Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: aesa
Record Dates: First submitted 2012-07-18; First posted 2012-07-23 (Estimated); Last update posted 2012-07-25 (Estimated); Status verified 2012-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Abraxane (Experimental): Abraxane for neoadjuvant chemotherapy
  Interventions: Drug: Abraxane

INTERVENTIONS:
Drug: Abraxane — Abraxane for neoadjuvant chemotherapy

SUMMARY:
Select 60 cases of women with breast cancer at clinical stage of T1-4N0-2M0. Then treat them with 4 cycles of TAC (Abraxane 260mg/m2,EPI 60 mg/m2 ,CTX 500 mg/m2, 21day/cycle) as neoadjuvant chemotherapy. Finally the investigators assess the efficacy and safety of Albumin-bound Paclitaxel.

DETAILED DESCRIPTION:
The investigators select 60 cases of women with breast cancer at clinical stage of T1-4N0-2M0. Then treat them with 4 cycles of TAC (Abraxane 260mg/m2,EPI 60 mg/m2 ,CTX 500 mg/m2, 21day/cycle) as neoadjuvant chemotherapy. Finally the investigators assess the efficacy and safety of Albumin-bound Paclitaxel.

ELIGIBILITY:
Inclusion Criteria:

1. Karnofsky ≥ 70
2. Provision of informed consent
3. Pathological confirmation of breast cancer
4. Tumor stage (TNM):T2-4bN0-3M0
5. Measurable disease as per RECIST criteria
6. Not previously treated with radiotherapy, chemotherapy or biological therapy.
7. Laboratory criteria:

   * PLT ≥ 100*109/L
   * WBC ≥ 4000/mm3
   * HGB ≥ 10g/dl
   * GOT,GPT,ALP ≤ 2*ULN
   * TBIL,DBIL,CCr ≤ 1.5*ULN

Exclusion Criteria:

1. Pregnant woman
2. History of organ transplantation
3. With mental disease
4. With severe infection or active gastrointestinal ulcers
5. With severe liver disease (such as cirrhosis), kidney disease, respiratory disease or diabetes
6. Disease-free period of other malignant tumor is less than 5 years (except cured basal cell skin cancer and cervical carcinoma in situ)
7. With heart disease
8. Experimental drug allergy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
therapeutic assessment | 6 months
  therapeutic assessment

SECONDARY OUTCOMES:
Adverse reactions and disease-free survival | 2 year
  Adverse reactions during the treatment and disease-free survival

OTHER OUTCOMES:
Recurrence or death | 5 years
  Recurrence or death

CONTACTS AND LOCATIONS:
Overall Officials: Jin Zhang, Professor, Study Chair — Tianjin Cancer Hospital
Locations (1):
- Tianjin Cancer Hospital, Tianjin, Tianjin Municipality, China